CLINICAL TRIAL: NCT06971874
Title: The Epidemiological Patterns of Obstructive Sleep Apnea Syndrome in Patients With Chronic Kidney Disease and Its Impact on Renal Prognosis
Brief Title: The Outcome of Chronic Kidney Disease Patients With Obstructive Sleep Apnea Syndrome
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-081
Record Dates: First submitted 2025-03-20; First posted 2025-05-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Diseases; OSAS (Obstructive Sleep Apneas Syndrome)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chronic kidney diseases with OSA
  Interventions: Other: No intervention
- chronic kidney diseases without OSA
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Obstructive sleep apnea (OSA) is highly prevalent in chronic kidney disease (CKD) patients and strongly linked to obesity, metabolic syndrome, and type 2 diabetes. Besides elevating cardiovascular disease risk, OSA may worsen renal function and diminish quality of life, making its understanding critical for CKD patient health.

This study will establish a large, long-term cohort of non-dialysis CKD patients to identify OSA risk factors, explore OSA's association with adverse renal outcomes, and determine OSA prevalence and epidemiological characteristics within the CKD population. The findings will provide a scientific foundation for early OSA identification, diagnosis, and intervention in CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign the informed consent form;

  * Aged ≥ 18 years and < 75 years;
  * Patients with CKD stages 3-4, with an eGFR of 15-60 ml/min/1.73m² calculated using the CKD-EPI formula for at least 3 months.

Exclusion Criteria:

* Patients receiving oxygen therapy or continuous positive airway pressure (CPAP) treatment;

  * Patients with other sleep disorders, including restless legs syndrome, periodic limb movement disorder, etc.;
  * Patients with other severe comorbidities: Severe heart failure (NYHA class III or IV); Myocardial infarction, unstable angina, or stroke within the past 3 months; Severe arrhythmias requiring medication or device therapy; Respiratory diseases, including COPD, asthma, thoracic deformities, etc.; Neurological disorders, including myasthenia gravis, Parkinson's disease, Alzheimer's disease, etc.; Active liver disease or severe hepatic insufficiency; Psychiatric conditions, including depression, anxiety disorders, etc.; History of malignancy within the past 5 years (except cured basal cell carcinoma); Uncontrolled hyperthyroidism;
  * Patients who underwent surgery or had acute infections within the past 3 months;
  * Current heavy alcohol consumption:Females: >3 drinks/day or >7 drinks/week; Males: >4 drinks/day or >14 drinks/week (1 standard drink = 14g of alcohol)
  * Current use of medications that may severely interfere with sleep, such as antipsychotics, antiepileptics, antiparkinsonian drugs, antidepressants, opioids, etc.;
  * Females who are pregnant or lactating at screening or baseline;
  * Inability to comply with the study due to: Low education level, language barriers, inability to tolerate or complete sleep monitoring, or other reasons preventing completion of study procedures (e.g., follow-up);
  * Deemed unsuitable for participation by the investigator's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The participants will be recruited from department of Nephrology, Nanfang Hospital
Sampling Method: Non-Probability Sample
Enrollment: 356 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The Progression of Chronic Kidney Diseases in CKD Patients | six months
  the progression of chronic kidney diseases is defined as: Patients had a 40% or a greater decrease in baseline eGFR(estimated Glomerular Filtration Rate); End-Stage Renal Disease (eGFR< 15 ml/min/1.73 m2, initiation of renal replacement therapy or renal transplantation )
Renal death or Cardiovascular death | six months
  Deaths Directly Caused by Renal or Cardiovascular Dysfunction or Their Acute or Chronic Complications

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events(MACE) | six months
  Composite endpoint including:
  Non-fatal myocardial infarction, Non-fatal stroke, Hospitalization due to unstable angina, heart failure, or transient ischemic attack (TIA), Cardiovascular (CV) death.
Cardiovascular Adverse Events | six months
  Individual components of the MACE composite endpoint.
24-hour urine protein(g/24h) | six months
  Total protein excreted in urine over 24 hours. Normal Range: <0.15 g/24h. Moderate proteinuria: >2.8 g/24h, suggestive of active glomerular disease.
Rate of eGFR Decline(mL/min/1.73m²/year) | six months
  Annualized decline in eGFR(estimated glomerular filtration rate). Decline Rate = Baseline eGFR - Follow-up eGFR. Normal decline rate: <-3 mL/min/1.73m²/year. Rate of eGFR Decline >5 mL/min/1.73m²/year indicating rapid progression.
Doubling of Serum Creatinine | six months
  A sustained ≥100% increase in serum creatinine(μmol/L) from baseline. Acute Kidney Injury: Occurring within 7 days. CKD progression: Over ≥3 months.
Cardiovascular Death | six months
  Death due to cardiovascular events
All-Cause Death | six months
  Death from any cause during the study period.
Apnea-Hypopnea Index (AHI) | 1 year
  Apnea: Complete cessation of airflow for ≥10 seconds. Hypopnea: Reduction in airflow by ≥30% accompanied by either ≥3% oxygen desaturation or an arousal (brief awakening).
  AHI = (Number of apneas + Number of hypopneas) / Total sleep hours. AHI for classifying the severity of sleep apnea. Mild Sleep Apnea: AHI 5-15 events/hour. Moderate Sleep Apnea: AHI 15-30 events/hour. Severe Sleep Apnea: AHI >30 events/hou.
Mean Blood Pressure(MBP, mmHg) | 1 year
  Average pressure in arteries during one cardiac cycle. Calculated from systolic and diastolic blood pressure. MBP=Diastolic BP+ 1/3*(Systolic BP-Diastolic BP). Approximately 70-100 mmHg (varies with age and health status).
Corrected QT Interval (QTc, ms) | 1 year
  Heart rate-adjusted duration of ventricular depolarization and repolarization. normal range:Adult males ≤440 ms;Adult females ≤460 ms. Significant Prolongation >480 ms (Regardless of gender).
left ventricular ejection fraction (LVEF, %) | 1 year
  Percentage of blood ejected from the left ventricle per heartbeat. Normal Range:55%-70% ; Mildly Reduced:41%-49%; Moderately Reduced:30%-40%; Severely Reduced:<30%.
Carotid Ultrasound Measurement Changes | 1 year
  Changes in carotid artery resistance index,carotid intima-media thickness (CIMT).
12-items Short-Form Healthy Survey Questionnaire (SF-12) | 1 year
  Assesses health-related quality of life across two dimensions:Physical Component Summary (PCS) and Mental Component Summary (MCS).
  Typical Range: Both PCS and MCS scores usually fall within 40-60 (mean ±1 standard deviation).
  Low score (<40) indicates worse physical or mental health; High score (>60) indicates strong physical or mental health.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China